CLINICAL TRIAL: NCT03141008
Title: Evaluation of Liver and Cardiometabolic Health Benefits on Low Carbohydrate Ketogenic Diet
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Obesity Treatment Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: HM20009338
Record Dates: First submitted 2017-04-18; First posted 2017-05-04 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Fatty Liver; Ketogenic Dieting
Keywords: Ketosis; NAFLD; Obesity
MeSH Terms: conditions — Obesity; Fatty Liver; Ketosis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — routine care labs will be done on patients including Comprehensive metabolic panel, A1c, lipids and insulin levels. Additional specimens will be taken for serum, urine, stool and saliva. These will be collected at time points 0, (additional timepoint of 1 month for saliva, stool and urine), 3 months, 6 months and 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ketogenic diet exposed group: Fibroscan changes with different diets:
  Patients in a weight loss program using a ketogenic diet. Will compare differences in Fibroscan and metabolic changes.
  Interventions: Other: Fibroscan changes with different diets
- NAFLD diet exposed group: Fibroscan changes with different diets:
  Patients in a NAFLD clinic using low calorie, low fat diet. Will compare differences in Fibroscan and metabolic changes.
  Interventions: Other: Fibroscan changes with different diets

INTERVENTIONS:
Other: Fibroscan changes with different diets — Observational study of liver fat and stiffness and cardiometabolic parameters comparing two different standard of care dietary regimens

SUMMARY:
To evaluate the impact of a Low Carbohydrate Ketogenic Diet (LCKD) weight loss program and compare to the standard of care program established for patients with Non-Alcoholic Fatty Liver Disease (NAFLD) on: (1) Liver fat and liver stiffness scores, (2) lipid profile and insulin sensitivity; and (3) depression scores and quality of life, and (4) Cardiometabolic measures such as cardiopulmonary exercise test (CPET) and transthoracic echocardiogram (TTE).

DETAILED DESCRIPTION:
This prospective pilot pragmatic trial will investigate the role of a LCKD weight loss program for obese patients (BMI ≥30 kg/m2) and compare it to the group of known obese NAFLD patients who receive dietetic counseling as part of their standard of care in a dedicated NAFLD program. All participants (n=50) will be recruited at Virginia Commonwealth University (VCU).

Patients will do initial paperwork including

Questionnaires QOL, eating disorder screen, depression screen:

QOL, eating disorder screen and depression screen.

Labwork:

Data will be collected from routine care labwork to include a fasting cholesterol panel, insulin, A1c and comprehensive panel (if they have not received these labs in the preceding 3 months), and at 6 and 12 months. A1c will be collected at 3,6,9 months as well (if A1c >/=7), or just additionally at 6 months if A1c <7

Study labs will be collected:

Blood at 0, 3, 6 and 12 months Urine, stool and saliva at 0, 1, 3 and 12 months

Fibroscan will be done at 0, 3, 6 and 12 months

Echo/CPET testing and Room calorimetry will be offered and the patients agreeing to do this will have them done at 0, 3 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria include patients aged 18 years and older, BMI ≥ 30, ALT (alanine transferase) > 19 (female) and > 30 (male) or radiographic evidence of hepatic parenchymal disease and seen in either the PIs weight loss clinic or a patient in the VCU NAFLD (non-alcoholic fatty liver disease) program.

Exclusion Criteria:

* Patients will be excluded if they have known other liver disease such as viral hepatitis, autoimmune hepatitis, liver transplant, severely ill, weekly alcohol use (>14 drinks in men and >7 drinks in women), HIV, pregnant females, those< 18 years, and prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 people from the PI's weight loss clinic using an a priori ketogenic diet. Will be compared with 50 people from a NAFLD clinic using a low calorie, low fat diet.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Change in liver fat and stiffness scores compared to control group as well as intrasubject trend | 0, 3, 6, 12 months
  Performed with a fibroscan

SECONDARY OUTCOMES:
Change in Cardiometabolic labs | 0, 6, 12 months (3 and 9 months for A1c if >7
  Lipids, A1c, Insulin, comprehensive metabolic panel
Other specialized testing | Only to a few of the eligible patients, 0, 3, 12 months
  Echo, cardiopulmonary exercise testing, room calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Susan Wolver, MD, Principal Investigator — VCU
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arulanandan A, Ang B, Bettencourt R, Hooker J, Behling C, Lin GY, Valasek MA, Ix JH, Schnabl B, Sirlin CB, Loomba R. Association Between Quantity of Liver Fat and Cardiovascular Risk in Patients With Nonalcoholic Fatty Liver Disease Independent of Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2015 Aug;13(8):1513-20.e1. doi: 10.1016/j.cgh.2015.01.027. Epub 2015 Feb 3. PMID 25661453
- [Background] Vanwagner LB, Bhave M, Te HS, Feinglass J, Alvarez L, Rinella ME. Patients transplanted for nonalcoholic steatohepatitis are at increased risk for postoperative cardiovascular events. Hepatology. 2012 Nov;56(5):1741-50. doi: 10.1002/hep.25855. PMID 22611040
- [Background] Francque SM, van der Graaff D, Kwanten WJ. Non-alcoholic fatty liver disease and cardiovascular risk: Pathophysiological mechanisms and implications. J Hepatol. 2016 Aug;65(2):425-43. doi: 10.1016/j.jhep.2016.04.005. Epub 2016 Jun 1. PMID 27091791
- [Background] Chang Y, Jung HS, Yun KE, Cho J, Cho YK, Ryu S. Cohort study of non-alcoholic fatty liver disease, NAFLD fibrosis score, and the risk of incident diabetes in a Korean population. Am J Gastroenterol. 2013 Dec;108(12):1861-8. doi: 10.1038/ajg.2013.349. Epub 2013 Oct 8. PMID 24100261
- [Background] Anstee QM, Targher G, Day CP. Progression of NAFLD to diabetes mellitus, cardiovascular disease or cirrhosis. Nat Rev Gastroenterol Hepatol. 2013 Jun;10(6):330-44. doi: 10.1038/nrgastro.2013.41. Epub 2013 Mar 19. PMID 23507799
- [Background] Ekstedt M, Hagstrom H, Nasr P, Fredrikson M, Stal P, Kechagias S, Hultcrantz R. Fibrosis stage is the strongest predictor for disease-specific mortality in NAFLD after up to 33 years of follow-up. Hepatology. 2015 May;61(5):1547-54. doi: 10.1002/hep.27368. Epub 2015 Mar 23. PMID 25125077
- [Background] Boursier J, Vergniol J, Guillet A, Hiriart JB, Lannes A, Le Bail B, Michalak S, Chermak F, Bertrais S, Foucher J, Oberti F, Charbonnier M, Fouchard-Hubert I, Rousselet MC, Cales P, de Ledinghen V. Diagnostic accuracy and prognostic significance of blood fibrosis tests and liver stiffness measurement by FibroScan in non-alcoholic fatty liver disease. J Hepatol. 2016 Sep;65(3):570-8. doi: 10.1016/j.jhep.2016.04.023. Epub 2016 May 2. PMID 27151181
- [Background] Wong RJ, Cheung R, Ahmed A. Nonalcoholic steatohepatitis is the most rapidly growing indication for liver transplantation in patients with hepatocellular carcinoma in the U.S. Hepatology. 2014 Jun;59(6):2188-95. doi: 10.1002/hep.26986. Epub 2014 Apr 25. PMID 24375711
- [Background] Prati D, Taioli E, Zanella A, Della Torre E, Butelli S, Del Vecchio E, Vianello L, Zanuso F, Mozzi F, Milani S, Conte D, Colombo M, Sirchia G. Updated definitions of healthy ranges for serum alanine aminotransferase levels. Ann Intern Med. 2002 Jul 2;137(1):1-10. doi: 10.7326/0003-4819-137-1-200207020-00006. PMID 12093239
- [Background] Targher G, Byrne CD, Lonardo A, Zoppini G, Barbui C. Non-alcoholic fatty liver disease and risk of incident cardiovascular disease: A meta-analysis. J Hepatol. 2016 Sep;65(3):589-600. doi: 10.1016/j.jhep.2016.05.013. Epub 2016 May 17. PMID 27212244
- [Background] Nagano M, Sasaki H, Kumagai S. Association of cardiorespiratory fitness with elevated hepatic enzyme and liver fat in Japanese patients with impaired glucose tolerance and type 2 diabetes mellitus. J Sports Sci Med. 2010 Sep 1;9(3):405-10. eCollection 2010. PMID 24149634
- [Result] Rinella ME. Nonalcoholic fatty liver disease: a systematic review. JAMA. 2015 Jun 9;313(22):2263-73. doi: 10.1001/jama.2015.5370. PMID 26057287